CLINICAL TRIAL: NCT00625469
Title: Treatment of Pulmonary Arterial Hypertension Secondary to Idiopathic Pulmonary Hypertension With Bosentan: A Single Center Pilot Study
Brief Title: Pulmonary Arterial Hypertension Secondary to Idiopathic Pulmonary Fibrosis and Treatment With Bosentan
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: competing studies did not allow enrollment
Sponsor: Rajan Saggar (Other)
Collaborators: Actelion (Industry)
Responsible Party: Sponsor-Investigator, Rajan Saggar, Principal Investigator, University of California, Los Angeles
Organization: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPF/PAH
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis
Keywords: pulmonary arterial hypertension; idiopathic pulmonary fibrosis; bosentan
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Idiopathic Pulmonary Fibrosis | interventions — Bosentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (3):
- treatment with bosentan (Experimental): patients with resting or exercise induced PAH receive bosentan in a randomized open label fashion
  Interventions: Drug: bosentan
- PAH group with no therapy (No Intervention): patients with resting or exercise PAH get randomized to receive no specific therapy
- No PAH and no therapy (No Intervention): patients with no evidence of either resting or exercise PAH receive no intervention but are followed until lung transplantation

INTERVENTIONS:
Drug: bosentan — 62.5mg orally bid for first month, followed by 125mg bid thereafter
  Other Names: tracleer
  Arms: treatment with bosentan

SUMMARY:
Pulmonary Arterial Hypertension (PAH) in the setting of Idiopathic Pulmonary Fibrosis(IPF)is a risk factor for morbidity and mortality in the peri-lung transplant(LT) setting. Currently there is no significant data to support the use of pulmonary vasodilators for PAH in the setting of interstitial lung disease such as IPF. The majority of IPF patients have PAH either at rest or during exercise. The study hypothesis is that bosentan may improve morbidity and mortality in the peri-LT setting in both IPF cohorts with either resting or exercise PAH.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate bosentan in the setting of exercise or resting pulmonary hypertension in patients with underlying pulmonary fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Pulmonary Fibrosis referred for lung transplantation
* Minimum 50 meter 6 minute walk distance
* No significant underlying liver disease

Exclusion Criteria:

* Significant liver disease or cirrhosis
* non ambulatory
* previous adverse reaction/allergy to Bosentan

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2009-06 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
6 minute walk distance | monthly assessement until date of lung transplantation
  ATS Guideline 6MW distance before and after intervention

SECONDARY OUTCOMES:
right heart catheterization hemodynamics | variable based on time between listing and actual lung transplantation
  pulmonary hemodynamics
chemokine peripheral blood analysis | monthly
  battery of chemokines analyzed from the peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Rajan Saggar, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - David Geffen School of Medicine UCLA, Los Angeles, California
  - Departments of Pulmonary and Critical Care, Cardiothoracic Surgery and Infectious Diseases at David Geffen School of Medicine at UCLA, Los Angeles, California